CLINICAL TRIAL: NCT02247960
Title: Antibiotic Prophylaxis for Urinary Catheter Removal After Radical Prostatectomy
Acronym: Abx
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis determined that the study should be concluded for futility.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jean Joseph, Professor of Urology and Oncology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSRB#50607
Record Dates: First submitted 2014-08-29; First posted 2014-09-25 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer; Urinary Tract Infection; Clostridium Difficile
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Tract Infections | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ciprofloxacin (Active Comparator): Antibiotic
  Interventions: Drug: Ciprofloxacin
- No Antibiotic (No Intervention): No Antibiotic

INTERVENTIONS:
Drug: Ciprofloxacin
  Other Names: Cipro
  Arms: Ciprofloxacin

SUMMARY:
The aim of this study is to determine whether antibiotics prophylaxis at the time of urinary catheter removal decreases the number of symptomatic urinary tract infections in patients after radical prostatectomy. In addition, the investigators aim to determine whether antibiotic prophylaxis is potentially harmful to patients (e.g. adverse reactions from antibiotic use, resistant bacteria in the urine, Clostridium difficile infections etc.). The investigators also aim to identify specific populations that may be at higher risk of developing urinary tract infections with urinary catheter use after radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will include patients undergoing radical prostatectomy for prostate cancer. Subjects will be randomized into control or treatment group.

Exclusion Criteria:

* Subjects with a history of adverse reaction to ciprofloxacin, or any other quinolone will be excluded. Subjects being treated with tizanidine or with a history of myasthenia gravis will be excluded. In addition, we will exclude patients with major immediate post-operative complications after prostatectomy including significant post-operative bleeding with known pelvic hematoma and known urine leak.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2014-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean V Joseph, M.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ciprofloxacin: Antibiotic
  Ciprofloxacin
Period: Patient Consent and Randomization
Arm/Group | Ciprofloxacin | No Antibiotic
Started | 85 | 90
Completed | 83 | 84
Not Completed | 2 | 6
Not completed — Physician Decision | 2 | 2
Not completed — Withdrawal by Subject | 0 | 4
Period: Catheter Removed
Arm/Group | Ciprofloxacin | No Antibiotic
Started | 83 | 84
Completed | 76 | 74
Not Completed | 7 | 10
Not completed — Lost to Follow-up | 7 | 10

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only collected on patients who had their catheter removed (ie. started period 2).
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciprofloxacin | No Antibiotic | Total
Number analyzed (Participants) | 83 | 84 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.49 (6.86) | 62.98 (6.82) | 62.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 83 | 84 | 167
Region of Enrollment [Number; unit: participants]
  United States | 83 | 84 | 167

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Positive Urinary Tract Infection
Description: After removal of the catheter, urine was tested for infection whenever symptoms were experienced by the participants from the time they enrolled to 12 months following their operation.
Time Frame: 12 months
Population: this outcome measure was only collected on patients who had their catheter removed (ie. started period 2)
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | No Antibiotic
Number analyzed (Participants) | 83 | 84
Participants | 5 | 5
Statistical Analysis 1: Comparison: Ciprofloxacin vs No Antibiotic; Test type: Superiority or Other; p = 1.00, Chi-squared

2. Secondary Outcome: Number of Participants Positive for Clostridium Difficile
Description: Development of Clostridium difficile was measured in stool for clostridium difficile infection by enzyme immunoassay (EIA) and/or polymerase chain reaction (PCR).
Time Frame: 3 months
Population: this outcome measure was only collected on patients who had their catheter removed (ie. started period 2)
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | No Antibiotic
Number analyzed (Participants) | 83 | 84
Participants | 0 | 3

3. Secondary Outcome: Number of Participants With Bacteria in Urine
Description: Bacterial cultures were performed on urine and the presence of the following bacteria was determined: Acinetobacter, Coagulase-negative staphylococci, Diptherioids, Escherichia coli, Enterobacter, Enterococcus, Klebsiella pneumonia, and Lactoferrin. Participants who were positive for one or more of these were considered positive.
Time Frame: 3 months
Population: 10 participants in the Ciprofloxacin arm and 16 participants in the no antibiotic arm did not have samples collected for testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | No Antibiotic
Number analyzed (Participants) | 73 | 84
Participants | 38 | 38

ADVERSE EVENTS:
Description: Adverse events were only collected on patients who had their catheter removed (ie. started period 2).
Arm/Group | Ciprofloxacin | No Antibiotic
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/84
Other Adverse Events (participants affected / at risk) | 0/83 | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes